CLINICAL TRIAL: NCT05518760
Title: A Multicenter Study to Assess the Effectiveness of an Inactivated COVID-19 Vaccine Against Hospitalized COVID-19
Brief Title: COVID-19 Effectiveness Study in the Philippines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of the Philippines (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); Mahidol Oxford Tropical Medicine Research Unit (Other); Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: SJREB-2021-103
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-12

CONDITIONS: COVID-19; Vaccine Effectiveness Against COVID-19; Hospitalized COVID-19
Keywords: COVID-19; Vaccine effectiveness; hospitalized COVID-19; inactivated COVID-19 vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Any remaining oropharyngeal and nasopharyngeal swab samples will be frozen at -70°C and will be kept at ICHHD-NIH-UPM for fifteen years. Consenting participants may rescind their consent at a later date and refuse the use of their samples (which will be destroyed) or data at any time up until the completion of the study. Future studies using the samples and data will undergo appropriate ethical reviews as required. Only the designated study personnel will have access to these specimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: A COVID-19 confirmed case is a patient with an acute respiratory illness and RT-PCR confirmation of SARS-CoV-2 infection (i.e. any positive RT-PCR results obtained prior to admission or after enrolment in the study). In case the patient has any inconsistent RT-PCR results (e.g. a positive followed by a negative or a negative followed by a positive result), he/s he/she will be considered as a COVID-19 confirmed case if he/she has at least one positive result during his/her illness under consideration.
  Interventions: Other: no intervention
- Test-negative control: A COVID-19 negative case is a patient with an acute respiratory illness, in whom all RT-PCR tests are negative for SARS-CoV-2
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
This is a multi-site, observational, prospective test negative design case-control study which primarily aims to determine the protective effectiveness of 2 doses of an inactivated COVID-19 vaccine at least 14 days after the second dose, against hospitalized virologically-confirmed SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Aged 18 years of age and above
* Residing in the catchment area of the participating hospital
* Admitted to the participating hospital with an acute respiratory illness
* Able and willing to provide a naso- and oro-pharyngeal swab for RT-PCR testing

Exclusion Criteria:

* 6.2.2.1 Refusal to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted for acute respiratory illness.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Number of hospitalized virologically-confirmed SARS-CoV-2 infection | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Deen, MD, MSc, Principal Investigator — ICHHD, University of the Philippines - National Institutes of Health; Michelle Ylade, MD, MSc, Principal Investigator — ICHHD, University of the Philippines - National Institutes of Health; Kristal An C Agrupis, MD, MSc, Principal Investigator — ICHHD, University of the Philippines - National Institutes of Health; Maria Vinna Crisostomo, MD, Principal Investigator — ICHHD, University of the Philippines - National Institutes of Health; Jedas Veronica Daag, RN, RMT, Principal Investigator — ICHHD, University of the Philippines - National Institutes of Health
Locations (1):
- Vicente Sotto Memorial Medical Center, Cebu City, Cebu Province, Philippines

IPD SHARING:
Plan to Share IPD: Undecided